CLINICAL TRIAL: NCT02675231
Title: monarcHER: A Phase 2, Randomized, Multicenter, 3-Arm, Open-Label Study to Compare the Efficacy of Abemaciclib Plus Trastuzumab With or Without Fulvestrant to Standard-of-Care Chemotherapy of Physician's Choice Plus Trastuzumab in Women With HR+, HER2+ Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Abemaciclib (LY2835219) in Women With HR+, HER2+ Locally Advanced or Metastatic Breast Cancer
Acronym: monarcHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15804; I3Y-MC-JPBZ (Other: Eli Lilly and Company); 2015-003400-24 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hormone Receptor Positive Breast Cancer; HER-2 Positive Breast Cancer
MeSH Terms: interventions — abemaciclib; Trastuzumab; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant (Experimental): 150 milligram (mg) abemaciclib given orally every 12 hours (Q12H) of a 21-day cycle; plus 8 milligram per kilogram (mg/kg) trastuzumab intravenous (IV) infusion on Day 1 of the cycle then a 6 mg/kg maintenance dose IV infusion on Day 1 of each subsequent cycle; plus 500 mg fulvestrant intramuscularly (IM) on day 1, 15 and 29 and then once every 4 weeks thereafter.
  Interventions: Drug: Abemaciclib; Drug: Trastuzumab; Drug: Fulvestrant
- 150 mg Abemaciclib + 8 mg/kg Trastuzumab (Experimental): 150 mg abemaciclib given orally Q12H of a 21-day cycle; plus 8 mg/kg trastuzumab IV infusion on Day 1 of the cycle then a 6 mg/kg maintenance dose IV infusion on Day 1 of each subsequent cycle.
  Interventions: Drug: Abemaciclib; Drug: Trastuzumab
- 8 mg/kg Trastuzumab + Standard of Care Chemotherapy (Active Comparator): 8 mg/kg trastuzumab IV infusion on Day 1 of a 21-day cycle then a 6 mg/kg maintenance dose IV infusion on Day 1 of each subsequent cycle plus standard of care single agent chemotherapy of physician's choice administered according to product label
  Interventions: Drug: Trastuzumab; Drug: Standard of Care Single Agent Chemotherapy

INTERVENTIONS:
Drug: Abemaciclib — Administered Orally
  Other Names: LY2835219
  Arms: 150 mg Abemaciclib + 8 mg/kg Trastuzumab; 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant
Drug: Trastuzumab — Administered IV
Drug: Fulvestrant — Administered IM
  Arms: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant
Drug: Standard of Care Single Agent Chemotherapy — Standard-of-care single-agent chemotherapy of physician's choice administered according to product label
  Arms: 8 mg/kg Trastuzumab + Standard of Care Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of abemaciclib plus trastuzumab with or without fulvestrant versus trastuzumab plus physicians choice standard of care chemotherapy in women with hormone receptor positive (HR+), human epidermal growth factor receptor 2 positive (HER2+) locally advanced or metastatic breast cancer after prior exposure to at least two HER2-directed therapies for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HR+, HER2+ breast cancer (BC)
* unresectable locally advanced recurrent BC or metastatic BC
* adequate tumor tissue available prior to randomization
* measurable and/or non-measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* previously received:

  * at least 2 HER2-directed therapies for advanced disease
  * participant must have received trastuzumab emtansine (T-DM1) in any disease setting
* must have received a taxane in any disease setting
* may have received any endocrine therapy (excluding fulvestrant)
* have postmenopausal status due to surgical / natural menopause or chemical ovarian suppression
* performance status (PS) of 0 to 1 on the Eastern Cooperative Oncology Group scale
* left ventricular ejection fraction (LVEF) of 50% or higher at baseline
* adequate organ function
* negative serum pregnancy test at baseline (within 14 days prior to randomization) and agree to use medically approved precautions to prevent pregnancy during the study and for 12 weeks following the last dose of abemaciclib if menopause induced by gonadotropin-releasing hormone (GnRH) agonist or radiation
* discontinued previous localized radiotherapy for palliative purposes or for lytic lesions at risk of fracture at least 2 weeks prior to randomization and recovered from the acute effects of therapy
* discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, and endocrine therapy), except trastuzumab, for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug, and recovered from the acute effects of therapy
* are able to swallow capsules

Exclusion Criteria:

* have visceral crisis
* known central nervous system (CNS) metastases that are untreated, symptomatic, or require steroids to control symptoms
* had major surgery within 14 days prior to randomization
* received prior treatment with any cyclin-dependent kinase (CDK) 4 and CDK 6 inhibitor
* received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of randomization for a nonmyelosuppressive or myelosuppressive agent, respectively
* have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study
* history within the last 6 months of symptomatic congestive heart failure, myocardial infarction, or unstable angina
* history within the last 12 months of any of the following conditions: syncope of cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest
* history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years
* active bacterial, fungal infection, or detectable viral infection
* have received any recent (within 28 days prior to randomization) live virus vaccination
* hypersensitivity to trastuzumab, murine proteins, fulvestrant, or to any of the excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (82):
- United States (30):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St Jude Medical Center, Fullerton, California
  - TRIO - Translational Research in Oncology-US, Inc., Los Angeles, California
  - USC Norris Cancer Hospital, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Care Associates Medical Group, Redondo Beach, California
  - Central Coast Medical Oncology Corporation, Santa Monica, California
  - Catholic Health Initiatives (CHI), Englewood, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - University of Miami Plantation, Plantation, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Winship Cancer Center Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - Fort Wayne Medical Oncology & Hematology, Inc., Fort Wayne, Indiana
  - St Joseph Cancer Center, Lexington, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Billings Clinic Research Center, Billings, Montana
  - Brookdale Hospital Medical Center, Brooklyn, New York
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Clinical Research Alliance, Inc, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Northwest Medical Specialties, PLLC, Puyallup, Washington
  - Swedish Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Argentina (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., CABA
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rioja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viedma
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kurralta Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleroi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - Universitair Ziekenhuis Leuven - Gasthuisberg, Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Namur
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - Instituto COI de Pesquisa Educação e Gestão, Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
  - Fundação Antonio Prudente - Hospital do Câncer A.C Camargo, São Paulo
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Newmarket
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ottawa
- France (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Cloud
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt am Main
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Achaia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sora
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., México
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badajoz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leicester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and european union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Tolaney SM, Goel S, Nadal J, Denys H, Borrego MR, Litchfield LM, Liu J, Appiah AK, Chen Y, Andre F. Overall Survival and Exploratory Biomarker Analyses of Abemaciclib plus Trastuzumab with or without Fulvestrant versus Trastuzumab plus Chemotherapy in HR+, HER2+ Metastatic Breast Cancer Patients. Clin Cancer Res. 2024 Jan 5;30(1):39-49. doi: 10.1158/1078-0432.CCR-23-1209. PMID 37906649
- [Derived] Tolaney SM, Wardley AM, Zambelli S, Hilton JF, Troso-Sandoval TA, Ricci F, Im SA, Kim SB, Johnston SR, Chan A, Goel S, Catron K, Chapman SC, Price GL, Yang Z, Gainford MC, Andre F. Abemaciclib plus trastuzumab with or without fulvestrant versus trastuzumab plus standard-of-care chemotherapy in women with hormone receptor-positive, HER2-positive advanced breast cancer (monarcHER): a randomised, open-label, phase 2 trial. Lancet Oncol. 2020 Jun;21(6):763-775. doi: 10.1016/S1470-2045(20)30112-1. Epub 2020 Apr 27. PMID 32353342
- See also: A Study of Abemaciclib (LY2835219) in Women With HR+, HER2+ Locally Advanced or Metastatic Breast Cancer (monarcHER) — https://trials.lilly.com/en-US/find/completed?trialname=%20I3Y-MC-JPBZ&externalRequestID=68cbce79-fbf1-46c5-852a-338ca6e2be85

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who either died due to any cause or were alive and on the study at the conclusion but off treatment.
Period: Overall Study
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Started | 79 | 79 | 79
Received at Least One Dose of Drug | 78 | 77 | 72
Completed | 74 | 71 | 74
Not Completed | 5 | 8 | 5
Not completed — Withdrawal by Subject | 2 | 4 | 2
Not completed — Lost to Follow-up | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant: 150 mg abemaciclib given orally every 12 hours (Q12H) of a 21-day cycle; plus 8 mg/kg trastuzumab intravenous (IV) infusion on Day 1 of the cycle then a 6 mg/kg maintenance dose IV infusion on Day 1 of each subsequent cycle; plus 500 mg fulvestrant intramuscularly (IM) on day 1, 15 and 29 and then once every 4 weeks thereafter.
- Total: Total of all reporting groups
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy | Total
Number analyzed (Participants) | 79 | 79 | 79 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.34 (10.25) | 54.99 (11.08) | 56.77 (12.37) | 55.37 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 79 | 237
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 12 | 37
  Not Hispanic or Latino | 58 | 52 | 56 | 166
  Unknown or Not Reported | 7 | 16 | 11 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 15 | 10 | 10 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 9
  White | 55 | 53 | 55 | 163
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 6 | 13 | 8 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 9 | 7 | 3 | 19
  United States | 20 | 8 | 17 | 45
  United Kingdom | 9 | 9 | 10 | 28
  Spain | 6 | 8 | 3 | 17
  Greece | 1 | 1 | 2 | 4
  Canada | 2 | 4 | 4 | 10
  South Korea | 11 | 9 | 10 | 30
  Belgium | 5 | 7 | 7 | 19
  Brazil | 3 | 1 | 4 | 8
  Italy | 2 | 5 | 2 | 9
  Mexico | 2 | 1 | 3 | 6
  Australia | 2 | 4 | 2 | 8
  France | 6 | 13 | 8 | 27
  Germany | 1 | 2 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS time was measured from the date of randomization to the date of investigator-determined objective progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Baseline to Progressive Disease or Death from Any Cause (Up To 36 Months)
Population: All enrolled participants. Censored participants: Abemaciclib + Trastuzumab + Fulvestrant=23; Abemaciclib + Trastuzumab = 18 and Trastuzumab + Standard of Care Chemotherapy = 27.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant: 150 mg abemaciclib given orally every 12 hours (Q12H) of a 21-day cycle; plus 8 mg/kg trastuzumab intravenous (IV) infusion on Day 1 of the cycle then a 6 mg/kg maintenance dose IV infusion on Day 1 of each subsequent cycle; plus 500mg fulvestrant intramuscularly (IM) on day 1, 15 and 29 and then once every 4 weeks thereafter.
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
Months | 8.3 [5.9 to 12.6] | 5.7 [4.2 to 7.2] | 5.7 [5.4 to 6.9]
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; PFS analysis was planned after approximately 165 PFS events occurred in the enrolled population, yielding greater than or equal to (≥) 80% power assuming a Hazard ration (HR) of 0·667 at an experiment-wise 2-sided alpha level of 0·2; Test type: Superiority — The abemaciclib plus trastuzumab plus fulvestrant arm will be compared to the standard of care (SOC) chemotherapy plus trastuzumab arm first, and the abemaciclib doublet arm will be compared to the SOC chemotherapy plus trastuzumab arm only if the test for the triplet vs the SOC chemotherapy plus trastuzumab arm is significant; p = 0.0506, Log Rank; Stratified by number of prior systemic regimens for advanced breast cancer (2 to 3 versus(vs) >3) and status of disease(measurable vs non-measurable)
Statistical Analysis 2: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7695, Log Rank; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With 1 Year Overall Survival (OS)
Description: OS is defined as the time from the date of randomization until death from any cause. For participants not known to have died by the data-inclusion cutoff date, OS is censored at the last date they were known to be alive. For each treatment arm OS rate at 1 year from the date of randomization was determined using the OS times and was estimated using the Kaplan-Meier method.
Time Frame: Randomization to date of death from any cause assessed at 1 year
Population: All randomized participants (including the censored participants). Number of participants censored were "150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant = 62," "150 mg Abemaciclib + 8 mg/kg Trastuzumab = 62," and "8 mg/kg Trastuzumab + Standard of Care Chemotherapy = 58."
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
percentage of participants | 77.2 [65.9 to 85.2] | 77.4 [66.1 to 85.3] | 69.8 [57.5 to 79.1]
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.241, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.36 to 1.30] — Stratified by the number of previous regimens (excluding single-agent endocrine therapy) for advanced breast cancer and the status of disease (measurable vs. non-measurable)
Statistical Analysis 2: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.313, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.38 to 1.36] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With 2 Year OS
Description: OS is defined as the time from the date of randomization until death from any cause. For participants not known to have died by the data-inclusion cutoff date, OS is censored at the last date they were known to be alive. For each treatment arm OS rate at 2 years from the date of randomization was determined using the OS times and was estimated using the Kaplan-Meier method.
Time Frame: Randomization to date of death from any cause assessed at 2 years
Population: All randomized participants (including the censored participants). Number of participants censored were "150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant = 47," "150 mg Abemaciclib + 8 mg/kg Trastuzumab = 47," and "8 mg/kg Trastuzumab + Standard of Care Chemotherapy = 41."
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
percentage of participants | 55.8 [43.5 to 66.4] | 55.7 [43.4 to 66.3] | 43.0 [30.9 to 54.5]
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.104, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.42 to 1.08] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.120, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.43 to 1.10] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With 3 Year OS
Description: OS is defined as the time from the date of randomization until death from any cause. For participants not known to have died by the data-inclusion cutoff date, OS is censored at the last date they were known to be alive. For each treatment arm OS rate at 3 years from the date of randomization was determined using the OS times and was estimated using the Kaplan-Meier method.
Time Frame: Randomization to date of death from any cause assessed at 3 years
Population: All randomized participants (including the censored participants). Number of participants censored were "150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant = 41," "150 mg Abemaciclib + 8 mg/kg Trastuzumab = 37," and "8 mg/kg Trastuzumab + Standard of Care Chemotherapy = 33."
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
percentage of participants | 46.7 [34.7 to 57.9] | 40.2 [28.6 to 51.5] | 29.9 [19.1 to 41.3]
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.049, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.42 to 1.00] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.153, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.48 to 1.12] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR): Objective Response Rate (ORR)
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Baseline to Objective Disease Progression (Up To 36 Months)
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
Percentage of participants | 32.9 [22.5 to 43.3] | 13.9 [6.3 to 21.6] | 13.9 [6.3 to 21.6]

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death from Any Cause (Up To 36 Months)
Population: All enrolled participants who received at least one dose of study drug and achieved CR or PR.Censored participants = 12 in 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant
  ; 3 participants in 150 mg Abemaciclib + 8 mg/kg Trastuzumab and 11 participants in 8 mg/kg Trastuzumab + Standard of Care Chemotherapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 26 | 11 | 11
Months | 12.5 [6.5 to 23.5] | 9.5 [2.8 to 22.7] | NA [4.1 to NA] — The median and upper limit of the 95% CI was not calculated due to the high censoring rate.

7. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR, PR, or Stable Disease (SD): Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Baseline to Objective Disease Progression (Up To 36 Months)
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
Percentage of participants | 78.5 [69.4 to 87.5] | 74.7 [65.1 to 84.3] | 67.1 [56.7 to 77.5]

8. Secondary Outcome: Percentage of Participants With Best Overall Response of CR, PR, or SD With Duration of SD for at Least 6 Months: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate defined as percentage of participants with best overall response of CR, PR, or SD with a duration of at least 6 months. CR, PR, or SD were defined using RECIST, v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. Percentage of participants = (participants with CR+PR+SD with a duration of at least 6 months /number of participants enrolled) *100.
Time Frame: Date of CR, PR or SD to 6 Months Post CR, PR or SD (Up To 36 Months)
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
Percentage of participants | 58.2 [47.4 to 69.1] | 45.6 [34.6 to 56.6] | 38.0 [27.3 to 48.7]

9. Secondary Outcome: Change From Baseline in Pain and Symptom Burden Assessment on the Modified Brief Pain Inventory-Short Form (mBPI-sf)
Description: The mBPI-sf is an 11-item instrument used as a multiple-item measure of cancer pain intensity. In addition to pain intensity (4 items), the mBPI-sf is designed for participants to record the presence of pain in general, pain relief, and pain interference with function (general activity, mood, ability to walk, ability to perform normal work, relations with others, sleep, enjoyment of life). Responses for the mBPI-sf items are captured through the use of 11-point numeric rating scales anchored at 0 (no pain or does not interfere) and 10 (pain as bad as you can imagine or completely interferes). The mBPI-sf recall period is 24 hours and typical completion time for this instrument is less than 5 minutes. Mean Interference Score data is reported here. Least square (LS) Mean value was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 36 Months)
Population: All enrolled participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 79 | 79 | 79
units on a scale | 0 (0.18) | 0.20 (0.18) | 0.31 (0.19)
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.232, MMRM Model — p-values are from Type 3 sums of squares mixed models repeated measures model (MMRM): Change from baseline = Treatment + Visit + Treatment*Visit + Baseline; Mean Difference (Final Values) = -0.31

10. Secondary Outcome: Change From Baseline in Symptom Burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, cognitive, emotional, and social), global health status, and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, higher scores represent a better level of functioning. For symptoms scales, higher scores represented a greater degree of symptoms. LS Mean value was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 36 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EORTC QLQ-C30 data for each EORTC QLQ-C30 items.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 72 | 72 | 69
units on a scale
  Global health status | -2.9 (1.6) | -5.9 (1.7) | -1.9 (1.8)
  Functional scale: Physical functioning | -1.0 (1.6) | -4.4 (1.6) | -4.5 (1.7)
  Functional scale: Role functioning | -2.7 (2.2) | -5.0 (2.3) | -8.2 (2.4)
  Functional scale: Emotional functioning: number analyzed (Participants) | 72 | 71 | 69
  Functional scale: Emotional functioning | 2.4 (1.7) | -0.4 (1.8) | 1.1 (1.8)
  Functional scale: Cognitive functioning | -1.8 (1.4) | -1.1 (1.5) | -1.6 (1.6)
  Functional scale: Social functioning: number analyzed (Participants) | 72 | 71 | 69
  Functional scale: Social functioning | -0.9 (1.9) | -0.9 (1.9) | -2.4 (2.0)
  Symptom scale: Fatigue | 1.8 (1.9) | 7.0 (2.0) | 4.7 (2.1)
  Symptom scale: Nausea and vomiting | 6.3 (1.4) | 5.6 (1.4) | 2.2 (1.5)
  Symptom scale: Pain | -2.5 (2.1) | 3.1 (2.1) | 4.3 (2.2)
  Symptom scale: Dyspnoea | 0.7 (1.9) | 2.9 (2.0) | 3.7 (2.1)
  Symptom scale: Insomnia | -4.4 (2.1) | -1.6 (2.2) | 2.0 (2.3)
  Symptom scale: Appetite loss | 6.3 (2.3) | 5.5 (2.4) | 2.4 (2.5)
  Symptom scale: Constipation: number analyzed (Participants) | 72 | 71 | 69
  Symptom scale: Constipation | -6.3 (1.9) | -10.5 (1.9) | -3.4 (2.0)
  Symptom scale: Diarrhoea | 21.5 (2.2) | 25.3 (2.3) | 2.2 (2.4)
  Symptom scale: Financial difficulties: number analyzed (Participants) | 72 | 71 | 68
  Symptom scale: Financial difficulties | 0.8 (2.0) | -1.9 (2.1) | -3.2 (2.2)
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Global health status; Test type: Superiority; p = 0.689, MMRM Model — [p-value comment as in outcome 9, analysis 1]; Least Square (LS) Mean Difference = -1.0, Standard Error of Mean 2.4
Statistical Analysis 2: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Functional scales: Physical functioning; Test type: Superiority; p = 0.141, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 3.4, Standard Error of Mean 2.3
Statistical Analysis 3: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Functional scale: Role functioning; Test type: Superiority; p = 0.095, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 5.5, Standard Error of Mean 3.3
Statistical Analysis 4: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Functional scale: Emotional functioning; Test type: Superiority; p = 0.591, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 1.3, Standard Error of Mean 2.5
Statistical Analysis 5: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Functional scale: Cognitive functioning; Test type: Superiority; p = 0.935, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -0.2, Standard Error of Mean 2.1
Statistical Analysis 6: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Functional scale: Social functioning; Test type: Superiority; p = 0.578, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 1.5, Standard Error of Mean 2.7
Statistical Analysis 7: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Fatigue; Test type: Superiority; p = 0.308, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -2.9, Standard Error of Mean 2.8
Statistical Analysis 8: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Nausea and vomiting; Test type: Superiority; p = 0.043, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 4.1, Standard Error of Mean 2.0
Statistical Analysis 9: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Pain; Test type: Superiority; p = 0.026, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -6.8, Standard Error of Mean 3.0
Statistical Analysis 10: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Dyspnoea; Test type: Superiority; p = 0.276, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -3.1, Standard Error of Mean 2.8
Statistical Analysis 11: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Insomnia; Test type: Superiority; p = 0.041, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -6.4, Standard Error of Mean 3.1
Statistical Analysis 12: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Appetite loss; Test type: Superiority; p = 0.262, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 3.9, Standard Error of Mean 3.4
Statistical Analysis 13: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Constipation; Test type: Superiority; p = 0.285, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -2.9, Standard Error of Mean 2.7
Statistical Analysis 14: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Diarrhoea; Test type: Superiority; p < 0.001, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 19.3, Standard Error of Mean 3.2
Statistical Analysis 15: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Symptom scale: Financial difficulties; Test type: Superiority; p = 0.180, MMRM Model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = 4.0, Standard Error of Mean 3.0

11. Secondary Outcome: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. Participants completed the 5-level (no problem, slight problem, moderate problem, severe problem, and inability or extreme problem), 5-dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) questionnaire concerning their current health state. Five dimensions of health status are each assessed with 5 response options and scored as a composite index which were anchored on a scale of 0 to 1 with a higher score representing better health status.LS Mean value was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 36 Months)
Population: All enrolled participants who received at least one dose of study drug with baseline and post-baseline EQ-5D 5L data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 72 | 72 | 68
units on a scale | 0.01 (0.02) | -0.01 (0.02) | -0.04 (0.02)
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.033, MMRM Model — p-values are from Type 3 sums of squares mixed models repeated measures model: Change from baseline = Treatment + Visit + Treatment*Visit + Baseline; LS Mean Difference = 0.05, Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.275, MMRM Model — [p-value comment as in outcome 11, analysis 1]; LS Mean Difference = 0.03, Standard Error of Mean 0.02

12. Secondary Outcome: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS)
Description: European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. The EQ-5D-5L is assessed using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine. A higher score indicates better health state. LS Mean value was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 36 Months)
Population: All enrolled participants who received at least one dose of study drug with baseline and post-baseline EQ-5D 5L VAS data.
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
Number analyzed (Participants) | 72 | 71 | 70
millimeter (mm) | 0.61 (1.4) | -1.64 (1.4) | -0.61 (1.5)
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.546, MMRM Model; LS Mean Difference = 1.22, Standard Error of Mean 2.02
Statistical Analysis 2: Comparison: 150 mg Abemaciclib + 8 mg/kg Trastuzumab vs 8 mg/kg Trastuzumab + Standard of Care Chemotherapy; Test type: Superiority; p = 0.620, MMRM Model; LS Mean Difference = -1.02, Standard Error of Mean 2.1

13. Secondary Outcome: Pharmacokinetics (PK): Minimum Steady State Concentration (Cmin,ss) of Abemaciclib and Its Metabolites (M2 and M20)
Description: Minimum Steady State Concentration (Cmin,ss) of Abemaciclib and Its Metabolites (M2 and M20) was evaluated. M2 and M20 are 2 major active metabolites of abemaciclib.
Time Frame: Cycle(C)1 Day(D)1,C1D15, C2D1, C2D8, C3D1,C3D15, C4D1, C5D1:pre-dose; C1D1, C2D1, C3D1, C4D1, C5D1:post-dose
Population: All enrolled participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab
Number analyzed (Participants) | 77 | 71
nanogram/milliliter (ng/mL)
  Abemaciclib | 134 (77) | 155 (53)
  M2 | 72.0 (120) | 96.5 (120)
  M20 | 136 (120) | 181 (130)

ADVERSE EVENTS:
Time Frame: Baseline till end of follow-up (Up to 6.5 years)
Description: All enrolled participants who received at least one dose of study drug.
Groups:
- 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant: 150 mg abemaciclib given orally every 12 hours (Q12H) of a 21-day cycle; plus 8mg/kg trastuzumab intravenous (IV) infusion on Day 1 of the cycle then a 6 mg/kg maintenance dose IV infusion on Day 1 of each subsequent cycle; plus 500mg fulvestrant intramuscularly (IM) on day 1, 15 and 29 and then once every 4 weeks thereafter.
Arm/Group | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant | 150 mg Abemaciclib + 8 mg/kg Trastuzumab | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy
All-Cause Mortality (participants affected / at risk) | 52/78 | 55/77 | 53/72
Serious Adverse Events (participants affected / at risk) | 24/78 | 15/77 | 14/72
Other Adverse Events (participants affected / at risk) | 76/78 | 75/77 | 68/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant (N=78) | 150 mg Abemaciclib + 8 mg/kg Trastuzumab (N=77) | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy (N=72)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 3 (5)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg Abemaciclib + 8 mg/kg Trastuzumab + 500 mg Fulvestrant (N=78) | 150 mg Abemaciclib + 8 mg/kg Trastuzumab (N=77) | 8 mg/kg Trastuzumab + Standard of Care Chemotherapy (N=72)
Anaemia (Blood and lymphatic system disorders) | 30 (47) | 20 (25) | 16 (19)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 18 (27) | 9 (13) | 10 (58)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 6 (7) | 4 (5) | 4 (16)
Neutropenia (Blood and lymphatic system disorders) | 38 (72) | 27 (59) | 26 (88)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (33) | 23 (42) | 5 (20)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (4) | 0 (0) | 1 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 3 (4) | 3 (3) | 1 (2)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Intraocular haematoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 7 (8) | 5 (5) | 2 (2)
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 4 (4) | 3 (3) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (9) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 24 (35) | 19 (26) | 16 (20)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (13) | 8 (9) | 15 (19)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 62 (169) | 60 (163) | 18 (33)
Dry mouth (Gastrointestinal disorders) | 4 (5) | 5 (6) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 8 (15) | 7 (8) | 6 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (5) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (6) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 38 (56) | 32 (48) | 26 (36)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 7 (9) | 8 (13)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (33) | 22 (27) | 11 (13)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2) | 1 (1)
Chills (General disorders) | 4 (5) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 45 (66) | 41 (57) | 32 (39)
Feeling of body temperature change (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gravitational oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 3 (3) | 6 (15) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 3 (4) | 1 (1) | 2 (2)
Malaise (General disorders) | 1 (1) | 3 (3) | 1 (1)
Mucosal dryness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 3 (4) | 4 (6)
Necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (7) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 4 (10) | 6 (9) | 7 (8)
Pain (General disorders) | 3 (3) | 2 (2) | 1 (2)
Peripheral swelling (General disorders) | 1 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 13 (18) | 5 (8) | 11 (17)
Swelling face (General disorders) | 1 (2) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Pseudocirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0) | 4 (5)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (6) | 5 (5) | 2 (2)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (5) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 2 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 12 (19) | 4 (5) | 8 (12)
Urinary tract infection (Infections and infestations) | 8 (16) | 10 (24) | 6 (9)
Vaginal infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Viral sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 3 (4) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (4)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (8) | 6 (9) | 8 (17)
Aspartate aminotransferase increased (Investigations) | 10 (11) | 7 (10) | 8 (22)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 7 (7) | 1 (1) | 2 (3)
Blood bilirubin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (5) | 2 (2) | 4 (8)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood chloride increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 10 (15) | 11 (14) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Cell marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 3 (4)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 3 (3) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Grip strength decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 6 (10) | 5 (5) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 19 (26) | 16 (20) | 13 (15)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 4 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6) | 3 (3) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (18) | 7 (14) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (21) | 12 (14) | 11 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (11) | 12 (14) | 6 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 7 (10)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 7 (8) | 10 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (6) | 8 (11)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7) | 10 (14) | 3 (3)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 4 (4) | 2 (4)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (19) | 11 (16) | 15 (18)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 5 (5) | 7 (8) | 15 (20)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1)
Abulia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3) | 5 (6)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 7 (9) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (9) | 5 (5)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (8) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (3) | 1 (2) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (31) | 12 (14) | 9 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 7 (9) | 13 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 7 (11) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 1 (1)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9) | 7 (8) | 8 (8)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 1 (1)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (4) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 13 (20)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (17) | 9 (9) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 15 (19) | 14 (20) | 9 (13)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Breast reconstruction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Nail operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Radiotherapy to brain (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (3)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 6 (9) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 3 (4) | 4 (6) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT02675231/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02675231/SAP_001.pdf